CLINICAL TRIAL: NCT00759850
Title: PaclitAxel or Sirolimus-Eluting Stent vs Bare Metal Stent in Primary Angioplasty (PASEO) Randomized Trial
Brief Title: Drug Eluting Stent (DES) in Primary Angioplasty
Acronym: PASEO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: San Giuseppe Moscati Hospital (Other)
Responsible Party: Emilio Di Lorenzo MD PhD, Division Of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM_DES01
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Drug Eluting Stent; Primary PCI
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Patient with ST elevation myocardial infarction randomly assigned to receive a Bare Metal Stent n=90)
  Interventions: Device: Drug Eluting Stent (DES)
- B (Experimental): Patient with ST elevation myocardial infarction randomly assigned to receive a Paclitaxel Eluting Stent (n=90)
  Interventions: Device: Drug Eluting Stent (DES)
- C (Experimental): Patient with ST elevation myocardial infarction randomly assigned to receive a Sirolimus Eluting Stent (n=90)
  Interventions: Device: Drug Eluting Stent (DES)

INTERVENTIONS:
Device: Drug Eluting Stent (DES) — Open-label randomization was performed after initial angiography by the treating physician when eligibility criteria were met. All patients received in the CCU 70U/Kg i.v. bolus of UFH plus 1000U/h infusion (to maintain an ACT of at least 200 seconds), aspirin intravenously (500 mg) and clopidogrel (300 mg loading dose). All patients received upstream Gp IIb-IIIa inhibitors administration as a routine adjunctive therapy before primary PCI. Postinterventional antiplatelet therapy for all patients included in the three study group, consisted of aspirin (100 mg) indefinitely and clopidogrel (75 mg for six months). Stenting procedures were performed according to standard techniques. The number and length of stents, and the type of BMS to be implanted, were left to the operator's discretion. The operator was allowed to implant DES to cover the entire length of the lesion with coverage of the entire stented segment and of 5 mm proximal and distal segments.
  Other Names: Primary Angioplasty; Cypher; Taxus

SUMMARY:
Stent implantation is the best treatment in patients with acute myocardial infarction (STEMI) referred for primary angioplasty (pPCI). However the occurrence of in stent restenosis is responsible for the need of repeat intervention. Both Sirolimus-eluting stents (SES) and Paclitaxel-eluting stents (PES) have been proven to virtually abolish in-stent restenosis in elective patients in simple e more complex lesions. Both SES and PES have raised concerns regarding occurrence of late stent thrombosis, especially in complex lesion subsets or in high risk patients. The PaclitAxel or Sirolimus-Eluting Stent vs Bare Metal Stent in primary angioplasty (PASEO) trial was a prospective, single-center, randomized trial evaluating the benefits of SES or PES as compared to BMS implantation in patients undergoing primary angioplasty for acute STEMI. From 1 October 2003 we randomized with 1:1:1 ratio, 270 patients with STEMI and treated with pPCI, to implantation of a bare metal stent (BMS n=90), PES (n=90) or SES (n=90).

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of STEMI, with initial onset of chest pain within the past 12 hours, an ECG demonstrating > 0.1 mV ST-segment elevation in 2 or more contiguous leads or documented new left bundle-branch block and were suitable candidates for percutaneous revascularization.

Exclusion Criteria:

* Active internal bleeding or a history of bleeding diathesis within the previous 30 days
* An history of intracranial hemorrhage
* Intracranial neoplasm
* Arteriovenous malformation or aneurysm
* Known allergy to sirolimus
* Paclitaxel
* Heparin, aspirin, or clopidogrel
* An history of stroke within 30 days or any history of hemorrhagic stroke
* History, symptoms, or findings suggestive of aortic dissection, fibrinolytic therapy within 24 hours
* History of thrombocytopenia, pregnancy, patients on warfarin or acenocoumarol within the last seven days
* Inability to obtain the informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2003-10; Primary Completion 2005-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary end point was target lesion revascularization (TLR) at 1-year follow-up | 1 year

SECONDARY OUTCOMES:
Cumulative combined incidence of death and/or reinfarction at 2 year; Cumulative incidence of in-stent thrombosis at 2 year; 3) Major Adverse Cardiac Events (MACE) (combined death and/or reinfarction and/or TLR) at 2 years | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Di Lorenzo, MD PhD, Principal Investigator — Division of Cardiology A.O. Moscati Avellino Italy
Locations (1):
- U.O. Cardiologia/UTIC, Avellino, Italy

REFERENCES:
- [Derived] Di Lorenzo E, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Mariello C, Siano F, Pagliuca MR, Stanco G, Rosato G, De Luca G. Benefits of drug-eluting stents as compared to bare metal stent in ST-segment elevation myocardial infarction: four year results of the PaclitAxel or Sirolimus-Eluting stent vs bare metal stent in primary angiOplasty (PASEO) randomized trial. Am Heart J. 2009 Oct;158(4):e43-50. doi: 10.1016/j.ahj.2009.03.016. PMID 19781402
- [Derived] Di Lorenzo E, De Luca G, Sauro R, Varricchio A, Capasso M, Lanzillo T, Manganelli F, Mariello C, Siano F, Pagliuca MR, Stanco G, Rosato G. The PASEO (PaclitAxel or Sirolimus-Eluting Stent Versus Bare Metal Stent in Primary Angioplasty) Randomized Trial. JACC Cardiovasc Interv. 2009 Jun;2(6):515-23. doi: 10.1016/j.jcin.2009.03.012. PMID 19539255